CLINICAL TRIAL: NCT04859907
Title: Bone Flap Fixation Systems For Craniotomy Procedures
Acronym: LOOP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NEOS Surgery (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NEO-LOO-2020-01
Record Dates: First submitted 2021-04-15; First posted 2021-04-26 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-02

CONDITIONS: Craniotomy
MeSH Terms: interventions — Bone Plates

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clamp-like system (Experimental)
  Interventions: Device: Clamp-like system
- Plates and screws (Active Comparator)
  Interventions: Device: Plates and screws

INTERVENTIONS:
Device: Clamp-like system — Craniotomy closure
  Other Names: Cranial LOOP
  Arms: Clamp-like system
Device: Plates and screws — Craniotomy closure
  Arms: Plates and screws

SUMMARY:
Clinical investigation to compare the clinical safety and performance of a clamp-like device for craniotomy closure, with the standard of care system, titanium plates and screws.

ELIGIBILITY:
Inclusion Criteria:

* The subject is 18 years or older.
* The subject can be implanted with the assigned craniotomy closure system according to its Instructions for Use.
* At least one post-operative medical image (CT scan or Magnetic Resonance image) is planned to be performed.
* Life expectancy higher than 6 months.
* The subject is willing to give his/her informed consent and to comply with the required follow-up.

Exclusion Criteria:

* The subject presents any of the contraindications of the assigned craniotomy closure system.
* Orbitozygomatic or mastoid craniotomies.
* Posterior fossa (skull base) surgeries.
* Combined used of craniotomy systems (plates and clamps).
* The subject is currently participating in an investigational drug or device study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-11-19 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Bone flap alignment score | 6 months
  1-4

SECONDARY OUTCOMES:
Frequency of adverse effects and device deficiencies (device safety) | 6 months
  Frequency and type of Device related Adverse effects (AE and SAE) and device deficiencies
Bone-flap alignment score | 0-7 days after surgery (before discharge)
  1-4
Surgeon usability questionnaire | 0 days after surgery
  Likert scale [1-7], where 1 is very difficult and 7 very easy
Device related artefacts in neuroimaging | 6 months
  frequency
Device-related bulges or visible offsets | 6 months
  frequency
Post-craniotomy headache | 6 months
  Incidence

CONTACTS AND LOCATIONS:
Locations (3):
- Maribor University Medical Center, Maribor, Slovenia
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario la Paz, Madrid